CLINICAL TRIAL: NCT00784914
Title: A Pilot Feasibility, Dose-Escalation Study Using Intracerebral Microdialysis to Assess the Neuropharmacodynamics of Temsirolimus in Patients With Primary or Metastatic Brain Tumors
Brief Title: A Feasibility, Dose-Escalation Study Using Intracerebral Microdialysis to Assess the Neuropharmacodynamics of Temsirolimus in Patients With Primary or Metastatic Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07064; P30CA033572 (NIH); CHNMC-07064; CDR0000617019 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-11-01; First posted 2008-11-04 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Brain and Central Nervous System Tumors; Metastatic Cancer
Keywords: adult anaplastic astrocytoma; adult diffuse astrocytoma; adult craniopharyngioma; adult choroid plexus tumor; adult brain stem glioma; tumors metastatic to brain; recurrent adult brain tumor; adult gliosarcoma; adult giant cell glioblastoma; adult ependymoblastoma; adult medulloblastoma; adult supratentorial primitive neuroectodermal tumor (PNET); adult anaplastic ependymoma; adult ependymoma; adult myxopapillary ependymoma; adult subependymoma; adult mixed glioma; meningeal melanocytoma; adult meningeal hemangiopericytoma; adult grade I meningioma; adult grade II meningioma; adult grade III meningioma; adult anaplastic oligodendroglioma; adult oligodendroglioma; adult pineoblastoma; adult pineocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neoplasm Metastasis; Astrocytoma; Craniopharyngioma; Choroid Plexus Neoplasms; Brain Neoplasms; Gliosarcoma; Glioblastoma; Neuroectodermal Tumors, Primitive; Medulloblastoma; Ependymoma; Glioma, Subependymal; Glioma; Meningioma; Oligodendroglioma; Pinealoma | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Active Comparator): Patients do not receive temsirolimus.
  Interventions: Other: cytokine levels
- Cohort 2 (Experimental): 48 hours after surgery, patients receive one 200 mg dose of temsirolimus IV.
  Interventions: Drug: temsirolimus; Other: pharmacological study; Other: cytokine levels

INTERVENTIONS:
Drug: temsirolimus — Receive temsirolimus IV
  Arms: Cohort 2
Other: pharmacological study — Plasma levels of temsirolimus and sirolimus will be evaluated in serial blood samples.
  Arms: Cohort 2
Other: cytokine levels — Dialysate samples are collected at regular intervals during the 96 hours following placement of the catheter to measure changes in levels of cytokines, chemokines and growth factors

SUMMARY:
RATIONALE: Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Studying samples of blood and tumor tissue from patients with cancer in the laboratory may help doctors learn more about how this treatment is used by the body.

PURPOSE: The purpose of this study is to evaluate the feasibility of using a microdialysis catheter to see what effect temsirolimus has on various biological substances associated with brain tumors over time.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of using a microdialysis catheter with a high cut-off membrane to perform neuropharmacodynamics (nPD) assessment of targeted therapy with a mammalian target of rapamycin (mTOR) inhibitor, where nPD is defined as changes in intracerebral levels of vascular endothelial growth factor (VEGF), interleukin-1ß (IL-1ß), and other cytokines.

Secondary

* Assess the relationship between temsirolimus dose and changes in intracerebral levels of VEGF, IL-1ß, and other cytokines.
* Compare changes in intracerebral cytokine levels to changes in systemic cytokine levels.
* Assess the relationship between the degree of microvascular proliferation and the tensin homologue deleted on chromosome 10 (PTEN) status in tumor tissue.
* Assess the relationship between changes in intracerebral cytokine levels after treatment with temsirolimus.

OUTLINE: Two cohorts of 6 patients will be enrolled in this study. All patients undergo debulking craniotomy or stereotactic biopsy and a placement of a intracerebral CMA 71 microdialysis (ICMD) catheter. Patients then are assigned to 1 of 2 treatment cohorts.

* Cohort 1: Patients do not receive temsirolimus. Dialysate samples will be collected at regular intervals during the 96 hours following placement of the catheter as well as serial blood samples to measure levels of cytokines, chemokines and growth factors that occur after neurosurgery.
* Cohort 2: Beginning 48 hours after surgery, patients receive a single 200 mg dose of temsirolimus IV. Dialysate samples will be collected at regular intervals during the 96 hours following placement of the catheter as well as serial blood samples to measure levels of cytokines, chemokines and growth factors that occur after neurosurgery. Plasma levels of temsirolimus and sirolimus will also be measured from the serial blood samples.

After completion of study therapy and removal of ICMD catheter, patients are followed for 30 days.

ELIGIBILITY:
Inclusion Criteria

Patients must be at least 18 years of age.

Patients must have either a primary or metastatic brain tumor(s).

Patients must be in need of a surgical debulking or a stereotactic biopsy for the purpose of diagnosis or differentiating between tumor progression and treatment-induced effects following radiation therapy + or - chemotherapy.

For patients in cohort 2, treatment with temsirolimus must not be contraindicated.

Patients in cohort 2 must not be taking any hepatic enzyme-inducing anticonvulsants (phenytoin, carbamazepine, phenobarbital, primidone, oxcarbazepine).

Patients who are taking strong CYP3A4 inducers or inhibitors such as clarithromycin, itraconazole, ketoconazole, nefazodone, telithromycin, rifampin, rifabutin, rifampacin, or St. John's Wort must discontinue the medication beginning at least one week prior to surgery and lasting for the duration of the study. The only exception will be dexamethasone which can be used post-operatively as indicated.

Patients must have a Karnofsky Performance Status >= 60% or an ECOG/Zubrod score of<= 2.

Patients must have recovered from any toxicity of any prior therapy.

Patients must have adequate bone marrow function (defined as an absolute neutrophil count of >= 1500 cells/mm3 and platelet count ≥ 100,000 cells/mm3), liver function with total bilirubin <= 2.0 mg/dl and AST (SGOT) <= 4 times the institutional upper limit of normal, and serum creatinine <=1.5 x the institutional upper limit of normal.

Patients must be able to understand and be willing to sign a written informed consent document.

The effects of temsirolimus on a developing fetus are unknown. Therefore, female patients of childbearing potential and sexually-active male patients must agree to use an effective method of contraception while participating in this study. Women of childbearing potential must have a negative pregnancy test <=2 weeks prior to registration.

Exclusion Criteria

Patients must not be planning to receive radiation, other chemotherapy or participate in another clinical trial from the time of surgery until the microdialysis catheters is removed.

Patients allergic to temsirolimus, sirolimus (rapamycin), or Dextran.

Patients with a coagulopathy, increased susceptibility to infection or bleeding disorders.

Patients on anticoagulant drug therapy.

Patients with uncontrolled diabetes.

Patients who have a serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.

Female patients who are pregnant or breast-feeding.

HIV-positive patients receiving anti-retroviral therapy are excluded from the study due to the possibility of PK interactions with temsirolimus; however, patients will not be routinely screened for HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of using a microdialysis catheter to assess the neuropharmacodynamics (nPD) of temsirolimus | Every 6 hours for 96 hours after confirmation that the microdialysis catheter is placed appropriately
Changes in intracerebral levels of vascular endothelial growth factor (VEGF), interleukin-1ß (IL-1ß), and other cytokines | Every 6 hours for 96 hours after confirmation that the microdialysis catheter is placed appropriately

SECONDARY OUTCOMES:
Relationship between temsirolimus dose and changes in intracerebral levels of VEGF, IL-1ß, and other cytokines | Every 6 hours for 96 hours after confirmation that the microdialysis catheter is placed appropriately
Relationship between the degree of microvascular proliferation and the tensin homologue deleted on chromosome 10 (PTEN) status in tumor tissue | 30 days after placement of the microdialysis catheter.
Relationship between changes in intracerebral cytokine levels after treatment with temsirolimus | Every 6 hours for 96 hours after confirmation that the microdialysis catheter is placed appropriately
Compare changes in intracerebral cytokine levels to changes in systemic cytokine levels. | Every 6 hours for 96 hours after confirmation that the microdialysis catheter is placed appropriately

CONTACTS AND LOCATIONS:
Overall Officials: Jana Portnow, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States